CLINICAL TRIAL: NCT00220909
Title: A Prospective, Randomized, Double-Blind Protocol to Compare the Efficacy of Lansoprazole to Ranitidine in Healing Pre-Existing and/or Preventing the Development of Gastroduodenal Stress Ulceration and Postoperative Bleeding in Patients Undergoing Elective Coronary Artery Bypass Graft or Cardiac Valve Replacement Surgery
Brief Title: Lansoprazole Preventing Gastroduodenal Stress Ulcerations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment slow
Sponsor: Temple University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TU4572
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Patients Undergoing Elective Coronary Artery Bypass Graft
Keywords: Gastric erosions; Proton pump inhibitors
MeSH Terms: interventions — Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole

SUMMARY:
The primary objective of this study is to determine whether lansoprazole, administered intravenously, can protect patients undergoing cardiac surgery from the development of and/or progression of previously undetected acid/peptic disorders (erosive esophagitis, gastric ulcer, duodenal ulcer, diffuse gastritis, duodenitis) as measured by the Lanza score and LA classification for esophageal injury.

The secondary objectives of this study are:

1. To determine if intravenous lansoprazole protects against the development of clinically important gastrointestinal bleeding in this population (overt bleeding or requiring blood transfusion).
2. To determine if intravenous lansoprazole maintains the intragastric pH above that for placebo throughout the study period.

DETAILED DESCRIPTION:
This is a randomized, double-blind single center study which compares the efficacy of lansoprazole by IV infusion daily (60 mg bolus followed by 6 mg per hour) compared to ranitidine 50 mg IV q12 h in healing pre-existing and preventing perioperative stress ulcers and associated upper GI bleeding.

Patients will undergo a complete history including a medication history for intake of ASA/NSAIDs/anticoagulants/antiplatelet agents, physical examination, complete blood count, complete metabolic profile, ECG's and chest x-rays which rule out an exclusionary illness. Female subjects will have a urine pregnancy test performed. They will then sign an informed consent to participate in this randomized, double-blind study protocol. Patients will be excluded if they are currently using acid suppressive therapy or if they have a history of gastric/duodenal ulcers or gastroesophageal reflux disease that has required acid suppressive therapy.

Patients will be randomized to receive either lansoprazole or ranitidine intravenously by continuous intravenous infusion on the morning of surgery and on each of the subsequent 4 days. Computer randomization will be used with the code kept by pharmacy. The allocation will be concealed. Medication will be delivered in a sealed, unlabeled container from the pharmacy. Patients will be stratified between placebo and lansoprazole by preceding ASA/NSAID use. Lansoprazole will be given as a 60 mg bolus preoperatively followed by 6 mg per hour throughout the duration of the study. At the time of airway intubation in the operating room for the surgery, a nasogastric tube with a built-in intragastric pH electrode (Zinetics, Inc) will be passed into the mid-stomach by the anesthesiologist in place of the standard nasogastric tube. Intragastric pH will be measured during the perisurgical period until the morning of postoperative day 4, 72 hours after surgery. At that time, the nasogastric tube/pH probe will be removed and patients will undergo esophagogastroduodenoscopy (EGD) under sedation with midazolam and fentanyl. During the endoscopy, the maximum number of submucosal hemorrhages and erosions in an endoscopic field from the anterior and posterior walls of the antrum will be counted. Modified Lanza scores for both the stomach and the duodenum will be determined to quantify gastric and duodenal erosions and ulcerations6. We will also determine the LA classification of esophageal injury and inflammation. Before removal of the endoscope, a wireless pH capsule (Bravo pH capsule; Medtronic, Inc) will be placed in the body of the stomach 12 cm below the squamocolumnar junction for an additional two day measurement of intragastric pH or until the time of discharge from the hospital if less than 48 hours from the EGD. Thus, intragastric pH will be monitored from the morning that the patient undergoes surgery for 6 days or until the time of discharge.

After completion of surgery, all patients will be followed with hemoglobin and hematocrit every 12 hours; all stools will be tested for blood qualitatively (Hemoccult) and quantitatively (Hemaquant). Postoperatively, hemoglobin level will be maintained at or above 10 gm% using packed red blood cell transfusions as needed. Transfusion requirements will be quantified. The times at which patients resume oral intake will be noted along with specific data on oral liquid and solid food composition.

ELIGIBILITY:
Patients with symptomatic coronary artery disease or valvular heart disease who require corrective cardiac surgery will be eligible to participate in this study.

Inclusion Criteria:

* Patients undergoing cardiovascular surgery, specifically elective coronary artery bypass graft or cardiac valve replacement surgery, at Temple University Hospital
* Able to provide informed consent

Exclusion Criteria:

* Evidence of active gastrointestinal bleeding
* Prior gastric (e.g. Billroth II) or esophageal surgery
* Pregnancy
* Pre-existing or current condition requiring acid-suppressive therapy - e.g. reflux esophagitis, gastric or duodenal ulcer
* Current use of acid-suppressive therapy, such as proton pump inhibitors or histamine type 2 receptor antagonists
* Contraindication to naso- or oro-gastric intubation (e.g. Zenker's diverticulum, esophageal stricture)
* Bleeding diathesis
* Allergy to lansoprazole
* Advanced renal disease (BUN>40 and/or creatinine>2.0.
* Advanced liver disease (Alkaline phosphatase, ALT, AST>2 x normal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Mucosal Erosions

SECONDARY OUTCOMES:
Blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fisher, MD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine, Philadelphia, Pennsylvania, United States